CLINICAL TRIAL: NCT06442670
Title: Understanding New Semantic Memory Learnings Across the Lifespan
Acronym: ULIS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-A00167-40
Record Dates: First submitted 2024-05-28; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-04

CONDITIONS: Neurodevelopmental Changes (Childhood, Ageing)
Keywords: Semantic memory; Childhood; Ageing; EEG
MeSH Terms: interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 6-7 years children
  Interventions: Device: Electroencephalography
- 10-11 years children
  Interventions: Device: Electroencephalography
- 20-35 years adults
  Interventions: Device: Electroencephalography
- 60-70 older adults
  Interventions: Device: Electroencephalography
- 70-80 older adults
  Interventions: Device: Electroencephalography

INTERVENTIONS:
Device: Electroencephalography — Phase synchrony during the completion of the semantic memory task

SUMMARY:
The aim of this research is to specify the changes in brain connectivity (i.e. EEG phase synchronisation between brain regions) associated with semantic learning between individuals belonging to different age groups.

DETAILED DESCRIPTION:
Semantic memory is a crucial concept in cognitive science. It has long been conceptualised as a static, amodal memory system containing knowledge about the world, concepts and symbols. Although recourse to this concept is inevitable, the mechanisms, both cognitive and neurobiological, that govern it are far from being elucidated. There are many debates and controversies in this fundamental field of cognitive science, and more specifically around the question of the acquisition and formation of knowledge in semantic memory. The literature on the development of semantic memory during ontogeny is full of contradictions.

A review of this literature highlights the many unanswered questions surrounding semantic memory. How quickly is information encoded and then consolidated into a format that justifies the term semantic knowledge? What are the neural bases underlying the formation of knowledge in semantic memory? How does semantic knowledge evolve through new episodes? How do these mechanisms evolve during ontogeny? To what extent can some semantic learning be preserved from cognitive ageing? In the face of these many questions, the literature highlights the lack of tasks enabling semantic memory to be approached in an operational manner and the need to specify the cerebral mechanisms involved at different ages of life.

The general hypotheses that will be tested as part of the ULIS project are as follows:

1. New semantic learning is possible independently of episodic memory processes.
2. This learning differs according to the age of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Non-opposition by the participant or those exercising parental authority in the case of minors
* French language fluency (assessed by the investigating team)
* Absence of global cognitive deficit attested by a score on the MOCA (Montreal Cognitive Assessment) scale greater than or equal to 26/30 (test carried out at inclusion).

Exclusion Criteria:

* Person subject to a guardianship, curatorship or safeguard of justice measure
* Non affiliation to a social security scheme

Ages: 6 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
EEG Phase synchrony differences between age groups | Through study completion, an average of 2 years

SECONDARY OUTCOMES:
Behavioral performance differences between age groups (semantic memory task) | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clémence Tomadesso, Study Chair — University Hospital, Caen

IPD SHARING:
Plan to Share IPD: Undecided